CLINICAL TRIAL: NCT04962399
Title: Association of Serum N/OFQ, IL-6 and IL-6 Gene Polymorphisms With Type 2 Diabetic Nephropathy
Brief Title: Relationship Between Serum N/OFQ and Type 2 Diabetic Nephropathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zheng Guo (Other)
Responsible Party: Sponsor-Investigator, Zheng Guo, professor, Second Hospital of Shanxi Medical University
Organization: Second Hospital of Shanxi Medical University (Other)
Other Study IDs: hanyi20210703
Record Dates: First submitted 2021-07-04; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Diabetic Nephropathy Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- DKD group: Patients with type 2 diabetes mellitus complicated with diabetic nephropathy diagnosed by the second hospital of Shanxi Medical University
  Interventions: Diagnostic Test: Enzyme linked immunosorbent assay
- TDM group: Type 2 diabetes mellitus without diabetic nephropathy
  Interventions: Diagnostic Test: Enzyme linked immunosorbent assay
- control group: Health examination population in the same period
  Interventions: Diagnostic Test: Enzyme linked immunosorbent assay

INTERVENTIONS:
Diagnostic Test: Enzyme linked immunosorbent assay — Serum N / OFQ and IL-6 levels were detected，and the genotype and allele frequencies of rs1800796 in IL-6 gene were determined.
  Other Names: Real time fluorescent quantitative PCR

SUMMARY:
At present, the early diagnosis ability of diabetic nephropathy (DKD) is relatively poor, leading to some missed diagnosis of early disease patients. At the same time, because DKD patients have complex metabolic disorders, once they develop to end-stage renal disease, compared with other renal diseases, the treatment of DKD is more difficult and the prognosis is poor. At present, the main treatment for DKD is to strengthen blood glucose control and control blood pressure through renin angiotensin aldosterone system (RAAS) to delay the occurrence and development of DKD, but it can not reduce the risk of most patients progressing to end-stage renal disease (ESRD). In recent years, it is becoming a new therapeutic target for DKD to control the inflammatory response by targeting the inflammatory factors and inflammatory signaling pathways. Therefore, this study attempts to explore the correlation between N / OFQ and the occurrence and development of type 2 DKD, and seek new theoretical basis for the potential treatment of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes patients are in line with the relevant diagnostic criteria in China's guideline for prevention and treatment of type 2 diabetes (2017 Edition).
* patients with diabetic nephropathy are in line with the relevant diagnostic criteria in the expert consensus on diabetic nephropathy (2014 Edition).

Exclusion Criteria:

* Primary kidney disease (e.g. acute and chronic glomerulonephritis, immune and hereditary nephropathy, pyelonephritis, gout related nephropathy, etc.)
* Abnormal changes of microalbuminuria and urine glucose caused by other factors (such as urinary system infection, fever, 24-hour strenuous exercise, intractable hypertension, congestive heart failure, pregnancy, ketoacidosis, etc.)
* Failure of other important organs (heart, lung and liver) in the whole body;
* Activity of urinary sediment;
* The glomerular filtration rate decreased by more than 30% within 2-3 months after treatment with angiotensin converting enzyme inhibitor (ACEI) or angiotensin Ⅱ receptor antagonist (ARB);
* Patients with cancer, trauma, stress and other endocrine diseases;
* Patients with type 1 diabetes and kidney injury;
* Congenital mental retardation or poor compliance;
* The informed consent was not signed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients in the second hospital of Shanxi Medical University from May 2021 to October 2022
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
N/OFQ | 24 hours
  Serum N / OFQ levels
IL-6 | 24 hours
  Serum IL-6 levels
rs1800796 | 24 hours
  The rs1800796 polymorphism in the promoter region of IL-6 gene was analyzed